CLINICAL TRIAL: NCT00348855
Title: Effects of a Series of Intensified Prevention Consultations on the Changes in Goals and Risk Factors in Hypertensive Patients at High Cardiovascular Risk
Brief Title: Study to Improve Quality of Care and Patient Health in the Field of Cardiovascular Risk Factors in General Practice
Acronym: ESCAPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collège National des Généralistes Enseignants (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Assistance Publique - Hôpitaux de Paris (Other); Laboratoires Takeda (Industry); Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Denis Pouchain, MD, Collège National des Généralistes Enseignants
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNGE20060702
Record Dates: First submitted 2006-07-03; First posted 2006-07-06 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: High Risk Hypertensive Patients
Keywords: High Blood Pressure; High cardiovascular risk; Type 2 diabetes; Reaching goals
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Compliance; Exercise; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention with one day training, electronic device to measure bood pressure, leaflet with goals and drug strategies according to guidelines, six specific cardiovascular consultations during two years, feed back on results of the intervention group at inclusion, year 1 and year 2.
  Specific consultations will be focused on goals to be reach, compliance, exercise and diet.
  Interventions: Other: Cardiovascular drugs strategies; Behavioral: Compliance; Behavioral: Exercise; Behavioral: Stop Smoking; Behavioral: Diet; Other: Feed Back
- 2 (No Intervention)

INTERVENTIONS:
Other: Cardiovascular drugs strategies — Implementation of drug strategies according to guidelines to try to reach goals proposed in these guidelines.
  Arms: 1
Behavioral: Compliance — Discussion about compliance and questionnaire to assess compliance at inclusion, Year 1 and Year 2.
  Arms: 1
Behavioral: Exercise — Discussion with the patient on necessity to have regular exercise. Assessment of exercise by questionnaire at inclusion, year 1 and year 2.
  Arms: 1
Behavioral: Stop Smoking — Minimal intervention
  Arms: 1
Behavioral: Diet — Discussion with the patient on his (her) alimentation during each of the six consultations and assessment of daily diet at inclusion, year 1 and year 2.
  Arms: 1
Other: Feed Back — Feed back on results in the intervention group at baseline, Year 1 ans Year 2.
  Arms: 1

SUMMARY:
Observational studies performed in France and abroad in hypertensive patients at high cardiovascular risk have shown a wide gap between the therapeutic targets reached in ambulatory patients and those set by guidelines. In primary prevention, in hypertensive patients at high cardiovascular risk (+ at least 2 risk factors), the gap is secondary to 1) the ignorance of the validated therapeutic targets and strategies, 2) the absence of global cardiovascular risk management, 3) the usual ambulatory medical practice, which is not adapted to a global cardiovascular prevention approach.

Objectives Principal. To demonstrate that a series of 5 specific prevention consultations over 2 years allows a greater number of hypertensive patients at high cardiovascular risk to reach the goals set by guidelines with no deterioration of their quality of life compared with no particular intervention.

Method Pragmatic, cluster-randomised controlled trial. At least 1904 high cardiovascular risk hypertensive patients will be included and followed up during two years by 268 teaching general practitioners from 23 regional teaching colleges. The regional teaching colleges will be randomised to avoid a contamination bias. The study will be coordinated by local coordinators at the college level.

Intervention In the intervention group, the investigators will have training, information, and feed back regarding the management of high risk hypertensive patients. The training will concern the targets to be reached, therapeutic strategies recommended by the AFSSAPS/HAS, and scientific data. The investigators will have an easy guide that can be used during consultations, and will be informed about tobacco withdrawal programs and education for improving diet, exercise and compliance.

In the control group, investigators will care for their patients as usual. End points Main: number of patients who reach all the therapeutic targets defined by the guidelines in the total study population, in the sub-group of patients with hypertension, but free of type-2 diabetes (T2D), and in the sub-group with hypertension and DT2.

Secondary: number of targets reached by the patients, changes in level of blood pressure, LDL-cholesterol, HbA1c, tobacco consumption, and use of aspirin if needed in the total population and its two subgroups, estimated cardiovascular risk, quality of life.

DETAILED DESCRIPTION:
Cluster randomised pragmatic controlled trial in general practice

ELIGIBILITY:
Inclusion Criteria:

* Treated High blood Pressure patients with at least two other cardiovascular risks

Exclusion Criteria:

* Secondary prevention

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1836 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of patients who reach all the therapeutic goals defined by the guidelines in the total study population, in the sub-group of patients with hypertension, but free of type-2 diabetes (T2D), and in the sub-group with hypertension and T2D. | At inclusion, year 1 and year 2

SECONDARY OUTCOMES:
Number of targets reached by the patients | At inclusion, year 1 and year 2
Quality of life measured with SF8 | At inclusion, year 1 and year 2
Compliance | At inclusion, year 1 and year 2
Exercise | At inclusion, year 1 and year 2
Diet | At inclusion, year 1 and year 2
Levels of blood pressure, LDL-Cholesterol, tobacco consumption in the whole population plus levels of HbA1c and aspirin use in the TD2 population | inclusion, year 1 and year 2

CONTACTS AND LOCATIONS:
Overall Officials: Denis POUCHAIN, MD, Principal Investigator — French National College of GP Teatchers; Michel LIEVRE, MD, Study Director — EZUS LYON; Dominique HUAS, MD, Study Director — French National College of GP Teatchers
Locations (2):
- France (2):
  - Service de Pharmacologie Clinique, Lyon
  - French National College of GP Teatchers, Vincennes

REFERENCES:
- [Derived] Lebeau JP, Cadwallader JS, Vaillant-Roussel H, Pouchain D, Yaouanc V, Aubin-Auger I, Mercier A, Rusch E, Remmen R, Vermeire E, Hendrickx K. General practitioners' justifications for therapeutic inertia in cardiovascular prevention: an empirically grounded typology. BMJ Open. 2016 May 13;6(5):e010639. doi: 10.1136/bmjopen-2015-010639. PMID 27178974
- [Derived] Pouchain D, Lievre M, Huas D, Lebeau JP, Renard V, Bruckert E, Girerd X, Boutitie F; French National College of Teachers in General Practice. Effects of a multifaceted intervention on cardiovascular risk factors in high-risk hypertensive patients: the ESCAPE trial, a pragmatic cluster randomized trial in general practice. Trials. 2013 Oct 1;14:318. doi: 10.1186/1745-6215-14-318. PMID 24083783
- See also: Related Info — http://www.cnge.fr